CLINICAL TRIAL: NCT00602004
Title: Early and Late Cardiac Effects of Arteriovenous Fistula Creation for Haemodialysis in End-stage Renal Failure and Their Possible Attenuation
Brief Title: Attenuation of Cardiac Effects of Arteriovenous Fistula Creation With Losartan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Melbourne Health (Other)
Responsible Party: Dr Anuradha Aggarwal, Royal Melbourne Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2006.059
Record Dates: First submitted 2007-03-08; First posted 2008-01-28 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Renal Failure; Left Ventricular Hypertrophy
Keywords: Arteriovenous fistula; hypertrophy; losartan
MeSH Terms: conditions — Renal Insufficiency; Hypertrophy, Left Ventricular; Arteriovenous Fistula; Hypertrophy | interventions — Losartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: losartan — losartan 50 mg a day

SUMMARY:
The primary objective is to determine if the use of losartan, an angiotensin II receptor blocker, can attenuate left ventricular hypertrophy, independent of its antihypertensive effects, in patients with near end stage chronic kidney disease (CKD) who have an arteriovenous fistula created.

Secondary outcomes include the impact of the medication on BNP and hyperkalaemia

DETAILED DESCRIPTION:
Study Design: This is a prospective double blind placebo control 2 arm, randomized (1:1) parallel group study in patients with near end stage renal failure who require creation of an arteriovenous fistula for future haemodialysis. Enrolment will be over a period of 12 months. The blinded phase will be for 3 months. The study design is summarized in Appendix 1. The study consists of a screening phase, a randomization phase and a treatment phase.

Patients will be randomized into 2 groups:

* Group 1 Losartan (50mg daily blinded) and 25 mg of atenolol
* Group 2 Placebo (blinded) and 25 mg of atenolol

Patients: Patients must comply with specified inclusion and exclusion criteria. The number of patients used will be sufficient to show a 15% difference in the left ventricular mass (LVM) between the two groups

Study Endpoints: The primary endpoint is the between group difference in LVM from baseline to 1 month.

Statistical Considerations: The analysis will be based upon an 'ANCOVA'-type linear regression model that includes baseline LVM and treatment group as explanatory variables, and final LVM as the outcome variable.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of CKD at near-end stage renal failure (CKD Stage IV) ( eGFR = 15-30 mls/min).
2. Age >18 years of age and <85 years of age.
3. Males and post-menopausal, sterile women. Non-pregnant pre-menopausal women should be on adequate contraception and have no intention of becoming pregnant during the duration of the study.
4. At baseline TTE LVEF>45%
5. Willing and able to give informed consent.

Exclusion Criteria:

1. Serum potassium level of more than 5.5 mmol/L
2. Acute myocardial infarction or cerebrovascular accident in the previous 6 months.
3. Severe uncontrolled hypertension (diastolic BP >100mmHg or systolic BP >160 mmHg)
4. Evidence or suspicion of renovascular disease.
5. Atrial fibrillation
6. Evidence or suspicion of collagen disease, cancer, psychiatric disorder that interferes with patient compliance, drug or alcohol abuse, pregnancy, breast feeding and ineffective contraception.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2006-10; Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
left ventricular hypertrophy | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Anuradha Aggarwal, Principal Investigator — Melbourne Health; Eugenia Pedagogos, FRACP,PhD, Principal Investigator — Melbourne Health
Locations (1):
- Royal Melbourne Hospital, Parkville, Australia

REFERENCES:
- [Derived] Zentner D, Pedagogos E, Yapanis A, Karapanagiotidis S, Kinghorn A, Alexiou A, Lee G, Raspudic M, Aggarwal A. Can losartan and blood pressure control peri arteriovenous fistula creation ameliorate the early associated left ventricular hypertrophic response a randomised placebo controlled trial. BMC Res Notes. 2012 May 29;5:260. doi: 10.1186/1756-0500-5-260. PMID 22642740